CLINICAL TRIAL: NCT02205385
Title: Targeted Reinnervation as a Means to Treat Neuromas Associated With Major Limb Amputation
Acronym: TMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gregory Dumanian, Professor of Surgery, Plastic and Reconstructive Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMR Neuroma; OR120021 (Other Grant/Funding Number: CDMRP, Department of Defense Peer Reviewed Orthopaedic Research Program)
Record Dates: First submitted 2014-07-23; First posted 2014-07-31 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Neuroma; Neuroma Amputation; Pain
Keywords: Neuroma; Amputee; Amputation Stump; Assessment, Pain
MeSH Terms: conditions — Neuroma; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Traction Neurectomy (Active Comparator): Patients will be randomized to either the current standard of care surgical treatment for neuromas (traction neurectomy) or the experimental intervention (targeted reinnervation). This arm involves the use of the current standard of care surgical treatment.
  Patients will undergo the same pre-operative evaluation, anesthesia, and dissection to identify the painful residual limb neuroma(s). In the active comparator arm, gentle traction will be applied to the nerve while excising the neuroma (traction neurectomy) allowing the nerve to retract more proximally. It may be buried in healthy muscle to further pad the nerve ending. The intention is to place the inevitable recurrent end-neuroma away from superficial locations in which it is likely to become mechanically irritated.
  Interventions: Procedure: Traction Neurectomy
- Targeted Muscle Reinnervation (Experimental): Patients will be randomized to either the current standard of care surgical treatment for neuromas (traction neurectomy) or the experimental intervention (targeted reinnervation). This arm involves the use of the experimental surgical treatment.
  Patients will undergo the same pre-operative evaluation, anesthesia, and dissection to identify the painful residual limb neuroma(s). Targeted muscle reinnervation involves transfer of residual nerves to otherwise redundant target muscles. Native motor innervation of the target muscle is cut, and the residual nerves-after excision of end-neuromas-are coapted to the motor end point of the motor nerve, close to its point of entry into the muscle.
  Interventions: Procedure: Targeted Muscle Reinnervation

INTERVENTIONS:
Procedure: Targeted Muscle Reinnervation
  Other Names: Targeted Reinnervation
  Arms: Targeted Muscle Reinnervation
Procedure: Traction Neurectomy
  Arms: Traditional Traction Neurectomy

SUMMARY:
Subjects are being asked to participate in this study because they have an arm or leg amputation and have developed pain related to a neuroma (an ongoing localized pain related to a cut nerve ending).

We are studying two different types of surgery to treat the neuroma pain. Today there are many surgical options reported which often means that there is no one best treatment. The surgery that shows the best success so far, involves cutting out the scarred nerve ending (neuroma) and burying the freshly cut nerve ending in a nearby muscle. Recently, a new surgery has been developed called targeted reinnervation (TR). This surgery connects these cut nerve endings to nerves going into nearby nonfunctional muscles. This surgery was developed to allow amputees to have better prosthesis control. By chance, neuroma pain improved significantly with TR. We, therefore, are conducting this clinical trial to evaluate which of these two surgeries best treats neuroma pain. We will ask all participants to fill out a questionnaire both before and after surgery. This will help us understand how a neuroma affects the quality of life of amputees and will allow us to understand which surgery leads to the best improvement in neuroma pain.

In order to confirm the presence and location of the neuroma before surgery, a magnetic resonance image (MRI) will be performed. Taking these pictures requires subjects to lie still for a short period of time but does not involve any invasive procedures. After surgery, the MRI will be done again, this time to see if the nerve shows signs of scarring.

DETAILED DESCRIPTION:
Loss of an arm or leg is a significant injury that affects a person's job prospects, personal relationships, and overall quality of life. Approximately 25% of all amputees will develop chronic local pain in the remaining part of their amputated limb. This pain is caused by neuromas- disorganized nerve endings and scar tissue that form when an injured nerve tries to heal. Every cut nerve will develop a neuroma unless the two ends of the nerve can be rejoined. With limb amputation, the nerves are cut and one end is lost with the limb, preventing the nerve from repairing itself. Instead, the cut nerve ending forms a painful neuroma. Chronic pain from neuromas is a major reason that amputees cannot wear or use their prostheses comfortably and increases their disability. The current standard surgical treatment for a neuroma is to cut if off and bury the nerve ending in a muscle, to provide cushioning when the neuroma grows back. Even though this is the best current treatment, it is not always successful.

Even when a limb is amputated, the nerves that used to control that limb still carry messages from the brain. Those messages are intended to tell the muscles how or when to move the missing limb, but after amputation, these limb-control nerves are no longer connected to muscles. In 2002, researchers at Northwestern Memorial Hospital in conjunction with the Rehabilitation Institute of Chicago developed a new type of surgery called targeted muscle reinnervation (TMR). In TMR, limb-control nerves are transferred so that they can control new target muscles. The neuromas from the limb-control nerves are removed, then the small nerve that controls the target muscle is cut. The two nerves are joined together so that the limb-control nerve can then grow into, or reinnervate the target muscle. After TMR, when the person tries to move the missing limb, the target muscle contracts instead and these signals can be detected and used to control a prosthesis. TMR has now been done successfully almost 100 times worldwide. Interestingly, almost all of the patients who had painful neuromas before TMR had no neuroma pain after surgery. This result was investigated in laboratory studies - both rat and rabbit amputee neuromas were "cured" with TMR. We think that giving the cut nerve endings somewhere to go and something to do prevents a neuroma from forming.

We plan to compare TMR versus the current standard surgical treatment for painful neuromas. We will measure the effectiveness of both surgeries using an internet-based amputee pain questionnaire. We will also use magnetic resolution imaging (MRI) to look at the nerves before and after surgery. We have received a grant to complete a 4 year study in four hospitals across the US, in around 200 patients, making this the largest neuroma study ever performed. We expect that TMR will be significantly more effective for neuroma pain than the standard treatment. This will change how patients with neuroma pain are treated and help thousands of patients with amputations.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18 years or older: the Patient Reported Outcomes Measurement Information System (PROMIS) questionnaire is not validated for pain-related evaluation in minors
* An upper limb amputation above the wrist with or without a residual limb or a lower limb amputation above the ankle with a residual limb (individuals with a hip disarticulation amputation lack suitable target muscles for TR)
* A neuroma within the residual limb: defined as patient-reported chronic localized pain consistent with a physical exam that demonstrates that the pain is related to a cut nerve and excludes other causes. There must be a supporting Tinel's sign on physical exam, MRI findings suggestive of a neuroma, or localization of a neuroma by prior intervention (surgical or otherwise) to distinguish the pain from phantom limb pain or cold intolerance that are nonspecific signs of nerve damage that would not be affected by treatment of a neuroma.
* English or Spanish speaking: the PROMIS questionnaire is available in English and parts are currently available in Spanish. The portions that are currently unavailable in Spanish will be translated into Spanish for the purposes of this study.

Exclusion Criteria:

* Prior TR Surgery: these patients have already had a procedure to improve their prosthetic function and in these cases the nerves have been shortened. To perform a second TR procedure with the previously shortened nerves would require a significant proximal dissection and potentially greater soft tissue morbidity than the standard treatment.
* Cognitive impairment, due to TBI or other causes, sufficient to adversely affect understanding of or compliance with study requirements, ability to respond to questionnaires, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant feedback through questionnaires is essential to this study.
* Pre-operative assessment that precludes the patient from being eligible for TR or control surgery due to technical surgical concerns.
* Significant other comorbidity: Any other medical issues or injuries that would preclude safe administration of anesthesia or surgical intervention.
* Participation in other ongoing studies related to neuropathic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Improvement in pain of the amputated limb after surgery | 12 months
  Difference in patient-reported pain scores before and after surgical treatment using the online survey tool.
  Compare patient-reported pre-operative survey results to those after surgical intervention at intervals over time (1 month, 3 months,6 months, 9 months,1 year, and then every six months thereafter until the conclusion of the study).

SECONDARY OUTCOMES:
Improvement in physical functioning, including prosthesis wear, after surgery | 12 months
  Using the same PROMIS platform, general health, physical functioning (including functional prosthesis wear), and satisfaction following surgery will also be assessed as important secondary outcomes, resulting in a more comprehensive and objective understanding of the effects of the two surgical approaches on neuroma pain.
  Another particularly useful tool for this study is the Orthotics and Prosthetics User Survey (OPUS) Functional Status. The OPUS is a validated instrument that assesses how well patients are using their prostheses. Thus, we will examine a very important secondary measure of neuroma pain-the ability to use a prosthesis. Prosthesis use is often the primary problem for individuals with painful neuromas; they hurt most during walking with a prosthesis or when wearing a prosthetic arm. Thus we expect OPUS to be a useful additional measure for quantifying the outcomes of the two types of neuroma surgeries
Using MRI as a tool to determine if targeted muscle reinnervation prevents neuroma recurrence | 1 year
  In our study, pre- and post-operative neuroma size (at one year) will be quantified using MRI scans. Pre-operative MRI measurements will be compared to the removed neuroma specimen to verify the accuracy of the modality. Post-operative MRI measurements will be used to assess whether a neuroma recurred at the site of the surgery and to determine the size of any new lesion.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center, San Antonio, Texas

REFERENCES:
- [Derived] Dumanian GA, Potter BK, Mioton LM, Ko JH, Cheesborough JE, Souza JM, Ertl WJ, Tintle SM, Nanos GP, Valerio IL, Kuiken TA, Apkarian AV, Porter K, Jordan SW. Targeted Muscle Reinnervation Treats Neuroma and Phantom Pain in Major Limb Amputees: A Randomized Clinical Trial. Ann Surg. 2019 Aug;270(2):238-246. doi: 10.1097/SLA.0000000000003088. PMID 30371518